CLINICAL TRIAL: NCT01480466
Title: Use of Electronic Health Records for Addressing Overweight and Obesity in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Heather J. Baer, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: K01HS019789 (AHRQ)
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Body mass index; Weight; Primary care
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obesity tools in electronic health record (Experimental): This arm will consist of a new set of tools within the electronic health record to help primary care clinicians address overweight and obesity with their patients.
  Interventions: Other: Obesity tools in the electronic health record
- Standard care (No Intervention): This arm is standard care for overweight/obesity.

INTERVENTIONS:
Other: Obesity tools in the electronic health record — The intervention is a set of new tools within the Partners electronic health record that are designed to assist primary care clinicians with the assessment and management of overweight and obesity in their patients.
  Arms: Obesity tools in electronic health record

SUMMARY:
Overweight and obesity are highly significant clinical and public health issues, affecting more than two-thirds of adults in this country; however, primary care clinicians often do not document overweight or obesity or discuss weight management with their patients. The objectives of the proposed research are to develop and evaluate a set of tools within electronic health records (EHRs) to assist primary care clinicians with the diagnosis and treatment of overweight and obesity and to help patients manage their weight.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (ages >= 20 years) who have a visit at a primary care practice at Brigham and Women's Hospital during the intervention period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65278 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
weight change over 6 months | Baseline, 6 months
  Change in weight from first visit during Stage 2 of intervention period until approximately 6 months later, among patients with BMI >= 25
weight change over 12 months | Baseline, 12 months
  Change in weight from first visit during Stage 2 of intervention period until approximately 12 months later, among patients with BMI >= 25

SECONDARY OUTCOMES:
Documentation of height | Baseline, 6 months, 12 months
  Percentage of patients with height recorded in the electronic health record
Documentation of weight | Baseline, 6 months, 12 months
  Percentage of patients with weight recorded in electronic health record within past year
Documentation of body mass index | Baseline, 6 months, 12 months
  Percentage of patients with body mass index calculated in electronic health record within past year
Diagnosis of overweight and obesity | Baseline, 6 months, 12 months
  Percentage of patients with BMI >= 25 with Overweight or Obesity on the Problem List in the electronic health record
Management of overweight and obesity | Baseline, 6 months, 12 months
  Percentage of patients with BMI >= 25 with evidence of treatment for overweight or obesity in the electronic health record

OTHER OUTCOMES:
Primary care clinician attitudes about management of overweight and obesity | baseline, 12 months
  Primary care clinician attitudes about management of overweight and obesity, assessed via an electronic survey
Patient attitudes and behaviors around weight management | baseline, 6 months
  Patient attitudes, beliefs, and behaviors around weight management (including diet, physical activity)

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Baer, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Baer HJ, Wee CC, DeVito K, Orav EJ, Frolkis JP, Williams DH, Wright A, Bates DW. Design of a cluster-randomized trial of electronic health record-based tools to address overweight and obesity in primary care. Clin Trials. 2015 Aug;12(4):374-83. doi: 10.1177/1740774515578132. Epub 2015 Mar 25. PMID 25810449